CLINICAL TRIAL: NCT01775228
Title: The Effect of a Professionally-guided Telephone Peer Support Intervention on
Brief Title: Effect of Peer Support Intervention on Early Recovery Outcomes Post Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Council of Cardiovascular Nurses (Other)
Responsible Party: Principal Investigator, Tracey JF Colella, RN, PhD, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 17897; UofC 17897 (Other: University of Calgary)
Record Dates: First submitted 2012-12-29; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Disease
Keywords: Depression, peer support, recovery, health services
MeSH Terms: conditions — Cardiovascular Diseases; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular follow up care (No Intervention): No intervention group - received routine follow up care following discharge from hospital after cardiac surgery (no peer support intervention).
- Peer Support intervention (Active Comparator): Support (informational, emotional and appraisal) in the form of like persons (i.e. age, gender) who have undergone CABG surgery with successful outcomes (post-recovery at least one year); peer support was provided by telephone for 6 weeks post cardiac surgery recovery.
  Interventions: Behavioral: Peer Support

INTERVENTIONS:
Behavioral: Peer Support — Support (informational, emotional and appraisal) in the form of like persons (i.e. age, gender) who have undergone CABG surgery with successful outcomes (post-recovery at least one year); peer support was provided by telephone for 6 weeks post cardiac surgery recovery.
  Other Names: Social Support
  Arms: Peer Support intervention

SUMMARY:
Recovery from coronary artery bypass graft (CABG) surgery is a complex process involving physical recuperation and psychological adjustment. The high prevalence of postoperative depression in this population may threaten optimal recovery. Peer support over the recovery period has promise to mitigate this threat. The purpose of this study was to examine the effect of a professionally-guided telephone peer support intervention on recovery outcomes including depression, social support and health care resource utilization.

In a randomized controlled trial, 185 male CABG surgery patients randomly assigned to an intervention (n=61) or usual care (n=124) group. Participants in the intervention group received weekly telephone calls from a peer volunteer over 6 weeks post discharge. At hospital discharge and at 6 and 12 weeks follow up, depression was measured using the Beck Depression Scale-II, social support was measured using the Shortened Social Support Scale and health care resource utilization was measured using items in the Postoperative Self Report of Recovery Questionnaire. Participants in the intervention group were also asked questions about their perceptions regarding peer support using the Peer Support Evaluation Inventory.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* > 35 years of age
* undergoing first-time traditional (sternotomy approach) CABG surgery
* an uncomplicated postoperative course
* standard length of hospital stay (four to eight days)
* had a telephone in the home
* able to hear telephone conversation.

Exclusion Criteria:

* had cardiac surgery procedures other than CABG surgery
* resided in a nursing home or long term care facility
* had any neurological or psychiatric disorder that may have impeded ability to self reflect or communicate
* had emergent cardiac surgery
* had sustained in-hospital post surgical complications of major significance (i.e., stroke, GI bleed, cardiac tamponade, renal failure, cardiac arrest, major sepsis of any origin, deep sternal wound infection, myocardial infarction with significant hemodynamic compromise)

Ages: 36 Years to 87 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Post operative depression | 6 weeks
  A disorder of mood characterized by sadness and loss of interest in usually satisfying activities, a negative view of the self and hopelessness, passivity, indecisiveness, suicidal ideations, loss of appetite, weight loss, sleep disturbances, and other physical symptoms. Some or all of these symptoms may be present, and depression can be categorized as mild, moderate, or severe/major according to scores measured on the Beck Depression Inventory II (BDI-II) (Diagnostic and Statistical Manual of Mental Health Disorders - Fourth Edition) (DSM-IV criteria).
Post operative depression | 12 weeks
  A disorder of mood characterized by sadness and loss of interest in usually satisfying activities, a negative view of the self and hopelessness, passivity, indecisiveness, suicidal ideations, loss of appetite, weight loss, sleep disturbances, and other physical symptoms. Some or all of these symptoms may be present, and depression can be categorized as mild, moderate, or severe/major according to scores measured on the Beck Depression Inventory II (BDI-II) (Diagnostic and Statistical Manual of Mental Health Disorders - Fourth Edition) (DSM-IV criteria).

SECONDARY OUTCOMES:
Perceptions of recovery | 6 and 12 weeks
  Includes biophysical recovery, return to activity, and return to social roles; perceptions focused on the absence or resolution of physiological and/or psychosocial clinical symptoms. (Perceptions of recovery were measured by the Postoperative Self-Report of Recovery Questionnaire (PSRRQ) over 12-weeks post-discharge.
Perceptions of social support | 6 and 12 weeks
  Resources provided by others that can take the form of emotional support, instrumental aid, information, and positive feedback as to one's importance, capabilities or self worth. Social support was measured using the Shortened Social Support Scale (SSSS).
Health services utilization | 6 and 12 weeks
  The consumption of health services (emergency room visits, regularly scheduled and unscheduled family physician visits and readmission to hospital) to meet health care needs as defined by the patient or the health care professional. This was measured by the number of health care visits/readmissions to hospital over 12-weeks post-discharge using the Postoperative Self Report of Recovery (PSRRQ).

OTHER OUTCOMES:
Perceptions of peer support | 12 weeks
  Evaluation of the different aspects of peer support received (supportive interactions, relationship qualities, perceived benefits, satisfactions with support received) as measured by the Peer Support Evaluation Inventory (PSEI).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn King, PhD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Background] Colella TJ, King KM. Peer support. An under-recognized resource in cardiac recovery. Eur J Cardiovasc Nurs. 2004 Sep;3(3):211-7. doi: 10.1016/j.ejcnurse.2004.04.001. PMID 15350230